CLINICAL TRIAL: NCT04556578
Title: Use of Extracorporeal CO2 Removal in Case of Moderate to Severe Acute Respiratory Distress Syndrome to Apply an Ultraprotective Mechanical Ventilation Strategy
Brief Title: Use of Extracorporeal CO2 Removal in Case of Moderate to Severe ARDS to Apply an Ultraprotective Mechanical Ventilation Strategy
Acronym: ECCO2R
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in current practice in intensive care, few inclusions achievable
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19-0548
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acue Respiratory Distress Syndrome
Keywords: ARDS; ECCO2R; Ultraprotective ventilation; Respiratory extracorporeal support; Mechanical power; Driving pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-flow ECCO2R (Experimental): Extracorporeal support using high flow circulation
  Interventions: Procedure: High-flow extracorporeal CO2 removal

INTERVENTIONS:
Procedure: High-flow extracorporeal CO2 removal — Applying of a CO2 removal using an extracorporeal circulation with a flow of 2-3.5L/min in order to reduce the aggression induced by the mechanical ventilation.

SUMMARY:
The extracorporeal CO2 removal (ECCO2R) has been recently proposed in case of Acute Respiratory Distress Syndrome (ARDS) in order to reduce pulmonary injuries induced by the mechanical ventilation. A reducing of tidal volume and/or respiratory rate is thus expected using this extracorporeal respiratory support. However, most of existing devices of ECCO2R can apply only a limited extracorporeal flow, often less than 1L/min, which limits the CO2 exchanges and does not allow to reach an ultraprotective ventilation. An extracorporeal flow higher should logically maximalize CO2 removal and allow reducing intensity of mechanical ventilation. Works focused on high-flow ECCO2R (2-3 L/min) in setting of ARDS are therefore mandatory to better understand apprehend the phenomena of gazes changes with this device and confirm the added-value in management of these specific patients.

DETAILED DESCRIPTION:
This is a prospective interventional study focused on a cohort population.

The included patients will be those affected by a severe ARDS (Berlin definition) requiring an aggressive mechanical ventilation and whom a high-flow ECCO2R was implemented.

The high-flow ECCO2R will be proposed in all patients with inclusions criteria with the 15 first days following their admission. The day of initiation of the high-flow ECCO2R will considered as Day 0 in our study.

A data collection will be focused on the respiratory parameters, clinical complications until ICU discharge and outcome, extracted from medical records.

The main endpoint will be the perrcentage of patients whom an ultraprotective ventilation could be applied successfully during more than 12h. Ultraprotective ventilation is defined in our work as follows: Tidal volume ≤ 3 mL/kg and respiratory rate ≤ 16/min associated with a PaCO2 ≤ 45mmHg and a PaO2 ≥ 55 mmHg.

The secondary endpoints will be durations of mechanical ventilation, ICU stay and hospitalization, as well as rheological behavior of extracorporeal circulation, respiratory parameters under high-flow ECCO2R, specific complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years old
* Patient suffering from ARDS including the 3 following parameters during more than 12 hours:

PaO2/FiO2 ≤200 Driving Pressure ≥15 cmH2O, Tidal Volume = 6 mL/kg PIT Respiratory rate ≥ 28/min

- Or patient hospitalized for severe bronchospasm or COPD exacerbation associating a persistent capnia ≥ 50 mmHg despite maximal mechanical ventilation (Vt = 6mL/kg PIT, respiratory rate ≥ 24/min)

Exclusion Criteria:

* Patients protected by law (Art.L 1121-5, 1121-6, 1121-8 du Code de la santé publique)
* Consent refusal from the patient or his/her next of kin and the impossibility to enrol using the emergency procedure
* Pregnant or breast feeding patient
* Absence of a French Health Care Insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
percentage of patient who obtained a safe ultraprotective ventilation | 12 hours
  a safe ultraprotective ventilation is defined by the four following parameters :
  1. Tidal Volume ≤ 3 mL/kg
  2. Respiratory Rate ≤ 16/min
  3. PaCO2 ≤ 45mmHg
  4. PaO2 ≥ 55 mmHg.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | up to Day 30
Hospital length of stay | up to Day 30
ICU length of stay | up to Day 30
Day 30 all-cause mortality | up to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
identified data used in the published manuscript will be shared in accordance with the applicable informed consent under which the data was collected
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.